CLINICAL TRIAL: NCT07108855
Title: Detection of Upper Gastrointestinal Tumour Depth and Demarcation by Quantified Fluorescence Molecular Endoscopy Using Systemic Administration of Indocyanine Green During Endoscopic Submucosal Dissection
Brief Title: Detection of Upper Gastrointestinal Tumour Depth and Demarcation Using Systemic Administration of Indocyanine Green During Endoscopic Submucosal Dissection
Acronym: BRIGHT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: METc 2025/002; NL88635.042.24 (Other: CCMO)
Record Dates: First submitted 2025-04-30; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Carcinoma; Gastric Carcinoma
Keywords: Indocyanine Green (ICG); Fluorescence Molecular Endoscopy
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic administration of ICG (Experimental): Indocyanine Green (ICG) will be administered systemically 30 minutes before endoscopic submucosal dissection (ESD). Near-infrared quantified fluorescence molecular endoscopy (qFME) will be performed during the procedure.
  Interventions: Drug: Indocyanine Green (IC-Green); Diagnostic Test: Fluorescence guided identification using indocyanine green

INTERVENTIONS:
Drug: Indocyanine Green (IC-Green) — Systemic administration of indocyanine green during the endoscopic procedure.
Diagnostic Test: Fluorescence guided identification using indocyanine green — Near-infrared quantified fluorescence molecular endoscopy (qFME) will be used during the endoscopic procedure.

SUMMARY:
Endoscopic submucosal dissection (ESD) is a relatively new technique to treat superficial cancers in the upper gastrointestinal (GI) tract. Previous studies reported high en bloc resection rates (95%-97%). However, R0 resection rates (84.5%) suggest that the tumour is not radically removed in all cases, resulting in a risk of tumour recurrence. One of the key challenges is the limited accuracy in determining the depth of cancer invasion. To reduce the risk of tumour recurrence, the endoscopist would greatly benefit from proper and complete visualization of the tumour margin and depth during ESD. Several studies have shown that near-infrared quantified fluorescence molecular endoscopy (qFME) could serve as a red flag detection method and might be a useful imaging tool for tumour demarcation in the upper GI tract. The aim of this study is to evaluate the feasibility of ICG-enhanced near-infrared qFME to determine tumour demarcation and tumour depth in upper GI tumours (e.g. superficial esophageal and/or gastric adenocarcinoma (T1)) during ESD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed superficial esophageal and/or gastric adenocarcinoma (T1) and are scheduled for ESD within the UMCG;
* Age of 18 years or older;
* Able to provide written informed consent.

Exclusion Criteria (contraindications for indocyanine green):

* Known allergy to indocyanine green;
* Known allergies to iodine, shellfish and/or clams;
* eGFR < 30 mL/min/1.73 m2;
* Pregnancy or breastfeeding;
* Hyperthyroidism.

  * Severe liver disease (ascites and cirrhosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of ICG-enhanced qFME to determine tumour demarcation and depth in upper gastrointestinal tumours during ESD | One week after the qFME procedure
  Feasibility will be assessed by analyzing the fluorescent imaging data obtained during and after the procedure. Visible fluorescence will be determined by calculating the target-to-background ratio (TBR), where the target is defined as the mean pixel intensity of the resection bed in areas displaying fluorescence.
Feasibility of ICG-enhanced qFME to determine tumour demarcation and depth in upper gastrointestinal tumours during ESD | One week after the qFME procedure
  Secondary evaluation will focus on whether visible fluorescence after resection correlates with an R1 resection grade based on histopathology.
Feasibility of ICG-enhanced qFME to determine tumour demarcation and depth in upper gastrointestinal tumours during ESD | After study completion, to be expected within 8 months
  Fluorescence will also be quantified using mucosal multi-diameter single-fiber reflectance / single-fiber fluorescence (MDSFR/SFF) spectroscopy, a non-invasive measurement technique.

SECONDARY OUTCOMES:
Visibility of the papilla of Vater and the intraduodenal part of the extrahepatic biliary anatomy by detecting fluorescent signal with ICG-enhanced qFME | One week after the qFME procedure
  Visibility is determined visual evaluation during the endoscopic procedure and calculating the TBR in the same manner as explained above.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No